CLINICAL TRIAL: NCT00443573
Title: Multicenter, Two-Stage Study to Evaluate the Safety and Efficacy of Second-Line Metastatic Colorectal Carcinoma Treatment With Recombinant NAPc2
Brief Title: Safety Study of Recombinant NAPc2 to Prevent Tumor Progression and Metastases in Metastatic Colon Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company suspended development of product.
Sponsor: ARCA Biopharma, Inc. (Industry)
Responsible Party: Ted Love, MD, Nuvelo, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAP-0601
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Colon Cancer
Keywords: metastatic colorectal carcinoma (mCRC); colorectal carcinoma (CRC); tissue factor; factor VIIa; rNAPc2; adenocarcinoma; targeted therapy; coagulation-dependent; RECIST; 5-FU-based chemotherapy; FOLFOX; FOLFIRI; leucovorin; XELOX
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Adenocarcinoma | interventions — Anticoagulants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: recombinant nematode anticoagulant protein c2 (rNAPc2) — escalating dose administered 2x/week sq.
  Other Names: anticoagulant

SUMMARY:
This is a multicenter, two-stage trial with the goal of evaluating up to 100 subjects. This trial will be performed to initiate identification of a safe and effective dose of twice-weekly, subcutaneous rNAPc2 for the second-line treatment of metastatic colorectal carcinoma in combination with contemporary 5-FU-based chemotherapy.

DETAILED DESCRIPTION:
Cytotoxic chemotherapy combining 5-fluorouracil and leucovorin with irinotecan (FOLFIRI) or oxaliplatin (FOLFOX) or, more recently, treatment with XELOX (Roche) (capecitabine + oxaliplatin) has been the main approach for the treatment of metastatic colorectal carcinoma (mCRC), but with the advent of targeted therapies, biologic treatments are becoming an area of intense interest. Tissue factor (TF) is a transmembrane glycoprotein expressed by upwards of 85% of mCRCs.

ELIGIBILITY:
* Tissue diagnosis of adenocarcinoma of the colon or rectum
* Documented metastatic disease with at least one measurable lesion by RECIST criteria
* Previously treated with 5-FU-based chemotherapy in the form of FOLFIRI, FOLFOX, or XELOX plus bevacizumab as first-line chemotherapy and have recorded progressive disease during treatment or after discontinuation of treatment, when discontinuation of treatment occurred less than 6 months before enrollment (Stage I) or randomization (Stage II)
* Estimated life expectancy of at least 6 months
* Age 18 to 75 years
* Last dose of adjuvant or radiosensitizing chemotherapy less than 6 months before enrollment
* No other active malignancy for which the subject is currently receiving treatment (other than mCRC)
* No ongoing therapy with or need for parenteral and oral antithrombotics including anticoagulants and anti-platelet agents (including aspirin) and thrombolytics
* No contraindication to systemic anticoagulation
* No contraindication to modified FOLFOX6 or FOLFIRI combination chemotherapy
* No receipt of any investigational compound within 28 days of enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
Safety measured by major hemorrhage (NCI CTCAE v3.0 grade 3 or greater), during and up to 30 days after completion of study drug administration or, if treatment is ongoing, by 8 months after study enrollment (Stage I) or randomization (Stage II) | 30 days after study completion

SECONDARY OUTCOMES:
Safety measured by adverse events | 30 days after study completion
Efficacy measured by new metastasis-free survival by 8 months | 8 months
Survival by 8 months | 8 months
Arterial or venous thrombosis | 8 months
Tumor response rate, as assessed by RECIST criteria | 30 days after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ted Love, MD, Study Chair — ARCA Biopharma, Inc.
Locations (1):
- LAC/USC Medical Center, Los Angeles, California, United States

REFERENCES:
- See also: Company Website — http://www.nuvelo.com